CLINICAL TRIAL: NCT03613233
Title: Quality of Life Assessment in Traditional and Microinvasive Glaucoma Surgery.
Brief Title: QoL Assessment in Traditional Glaucoma Surgery and MIGS.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Marek Rekas, płk prof. Marek RĘKAS, MD, PhD, Military Institute od Medicine National Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0000000417
Record Dates: First submitted 2018-06-29; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Glaucoma
Keywords: MIGS; canaloplasty; glaucoma; glaucoma surgery; glaucoma implant; deep sclerectomy; iridencleisis; QoL; quality of life; NEI VFQ 25
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional glaucoma surgery (Active Comparator): glaucoma procedures such as trabeculectomy, iridencleisis, non - penetrating deep sclerectomy
  Interventions: Procedure: Glaucoma surgery
- microinvasive glaucoma surgery (MIGS) (Active Comparator): glaucoma procedures such as : canaloplasty (traditional, ABiC, modified), iStent, XEN, Cypass,Hydrus- and with any other microinvasive IOP reducing device
  Interventions: Procedure: Glaucoma surgery

INTERVENTIONS:
Procedure: Glaucoma surgery — phacoemulsification
  Other Names: cataract surgery when required

SUMMARY:
Quality of Life assessment before and after various glaucoma surgery (traditional and microinvasive (MIGS)).

DETAILED DESCRIPTION:
Patients qualified for glaucoma surgical procedure fill in QoL questionnaire (NEI VFQ 25) at baseline (pre-operatively) and 3 months after glaucoma surgery. Additional data will be collected such as demographic data and medical data, visual acuity, intraocular pressure, number of glaucoma medications, stage of glaucoma based on visual field assessment, medical ophthalmic history, intra and postoperative complications, postoperative interventions.

ELIGIBILITY:
Inclusion Criteria:

patients qualified for glaucoma surgery in Military Institute of Medicine - based on following Inclusion Criteria:

* all glaucoma types with characteristic glaucoma changes (biomicroscopic ,visual field) with documented glaucoma progression
* patients not tolerating antiglaucoma medications,
* patients with poor compliance
* progression in visual field

Exclusion Criteria:

* active inflammatory disease
* pregnancy
* mental disease or emotional instability
* general steroid therapy
* inability to fill in the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
NEI VFQ 25 quality of life score change | baseline (0-30 days; pre-operative) and three months after surgery
  NEI VFQ 25 baseline and 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Military Institute of Medicine, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided